CLINICAL TRIAL: NCT04645043
Title: The Effect of Real Time Ultrasound Guided Esophageal Pressure on Preventing Gastric Insufflation in Infants and Children: an Exploratory Study
Brief Title: Ultrasound Guided Esophageal Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009-150-1160
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Aspiration; Infant Conditions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- US_Eso (Experimental): US application on the participant
  Interventions: Other: US_Eso

INTERVENTIONS:
Other: US_Eso — After applying ultrasound guided esophageal pressure, the peak inspiratory pressure increased from 10cmH2O to 24cmH2O (increased by 2 cmH2O) during mask ventilation.

SUMMARY:
The investigator aimed to evaluate the effect of ultrasound guided esophageal pressure on the incidence of gastric insufflation during anesthetic induction in infants and small children undergoing general anesthesia.

DETAILED DESCRIPTION:
effect of ultrasound guided esophageal pressure on the incidence of gastric insufflation in children

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia with endotracheal intubation

Exclusion Criteria:

* patients with hypertrophic pyloric stenosis
* patients with delayed gastric emptying
* patients with esophageal stenosis
* patients with at risk of gastric aspiration
* patients with ileus, hepatomegaly, ascites (cannot visualize gastric antrum with ultrasound)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
the incidence of gastric air insufflation | during face mask ventilation, maximum 3 minutes.
  the incidence of gastric air insufflation during induction of anesthesia when applying real time ultrasound guided esophageal pressure.

SECONDARY OUTCOMES:
Gastric insufflation detected by esophageal ultrasound | during face mask ventilation, maximum 3 minutes.
ventilatory parameters | during face mask ventilation, maximum 3 minutes.
  tidal volume, end tidal carbon dioxide, minimal oxygen saturation
POGO (percentage of glottic opening) score | during endotracheal intubation, maximum 3 minutes
  POGO (percentage of glottic opening, 0-100) score with videolaryngoscope
relative position of esophagus with trachea | during anesthetic induction, maximal 3 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, Soul-t'ukpyolsi, South Korea

REFERENCES:
- [Derived] Kim EH, Cho SA, Kang P, Song IS, Ji SH, Jang YE, Lee JH, Kim JT, Kim HS. Ultrasound-guided esophageal compression during mask ventilation in small children: a prospective observational study. BMC Anesthesiol. 2022 Aug 15;22(1):257. doi: 10.1186/s12871-022-01803-5. PMID 35971064